CLINICAL TRIAL: NCT07042204
Title: Effectiveness of Extended Platelet-Rich Fibrin (ePRF) Alone and in Combination With Bioactive Glass Nanoparticles in the Treatment of Grade II Furcation Defects
Brief Title: Effectiveness of E-prf Alone and in Combination With Bioactive Glass Nanoparticles in Grade II Furcation Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merna Nasser Mohamed Mostafa Ibrahim Elnahas (Other)
Responsible Party: Sponsor-Investigator, Merna Nasser Mohamed Mostafa Ibrahim Elnahas, BDS, Clinical demonstrator, Oral Medicine, Periodontology, Diagnosis and Oral Radiology Department, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A03011023OM
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): 10 grade II furcation defects will be treated by extended platelet-rich fibrin (ePRF) alone.
  Interventions: Procedure: Group I (extended platelet-rich fibrin)
- Group II (Experimental): 10 grade II furcation defects will be treated by bioactive glass nanoparticles mixed with extended platelet-rich fibrin (BGn+ePRF).
  Interventions: Procedure: Group II (bioactive glass nanoparticles mixed with extended platelet-rich fibrin)
- Group III (Active Comparator): 10 grade II furcation defects will be treated by bioactive glass nanoparticles with collagen membrane.
  Interventions: Procedure: Group III (bioactive glass nanoparticles and covered by a collagen membrane)

INTERVENTIONS:
Procedure: Group I (extended platelet-rich fibrin) — mucoperiosteal flap will be raised through sulcular incisions Debridement of granulation tissue from the osseous defect and furcation will be filled with (ePRF) at the first group
  Arms: Group I
Procedure: Group II (bioactive glass nanoparticles mixed with extended platelet-rich fibrin) — bioactive glass nanoparticles mixed with extended platelet-rich fibrin (BGn+ePRF)
  Arms: Group II
Procedure: Group III (bioactive glass nanoparticles and covered by a collagen membrane) — bioactive glass nanoparticles and covered by a collagen membrane
  Arms: Group III

SUMMARY:
The aim of the study is to evaluate and compare the effectiveness of extended platelet-rich fibrin (ePRF) alone and in combination with bioactive glass nanoparticles in the treatment of grade II furcation defects clinically and radiographically.

DETAILED DESCRIPTION:
A total of 30 grade II furcation defects will be randomly divided into three groups as follows:

Group I: 10 grade II furcation defects will be treated by extended platelet-rich fibrin (ePRF) alone.

Group II: 10 grade II furcation defects will be treated by bioactive glass nanoparticles mixed with extended platelet-rich fibrin (BGn+ePRF).

Group III: 10 grade II furcation defects will be treated by bioactive glass nanoparticles with collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Glickman's grade II furcation defects in molars probing depth (PD) ≥5 mm horizontal PD ≥3 mm.
* The patients are in good systemic health and had not undergone any periodontal surgery in the areas to be treated within the prior 12 months.

Exclusion Criteria:

* Smokers and tobacco chewers.
* Patients that take any medications within the past 6 months that could alter their periodontal status.
* pregnant or lactating females.
* Patients with known allergy to materials or drugs that will be used or prescribed in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-08-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the amount of bone fill vertically and horizontally obtained in the treatment of grade II furcation defects calculated from CBCT data in millimeters | 6 months follow up

SECONDARY OUTCOMES:
the secondary outcomes include improvements (decrease)of probing depth in millimetres | 3 and 6 months follow up
  Using UNC-15 periodontal probe to measure the probing depth from the base of the pocket to the free gingival margin. All measurements will be rounded off to the nearest millimetre.
the secondary outcomes include improvements (decrease)of clinical attachment level loss in millimetres | 3 and 6 months follow up
  using a UNC-15 periodontal probe to measure clinical attachment level loss from the cemento-enamel junction (CEJ) to the pocket depth. All measurements will be rounded off to the nearest millimetre
the secondary outcomes include improvements (decrease) of gingival recession measured in millimetres | 3 and 6 months follow up
  Using a UNC-15 periodontal probe to measure gingival recession from cemento-enamel junction (CEJ) to the free gingival margin. All measurements will be rounded off to the nearest millimetre
the secondary outcomes include improvements (decrease) of gingival bleeding index | 3 and 6 months follow up
  It's performed through gentle probing of the orifice of the gingival crevice using a UNC-15 periodontal probe. If bleeding occurs within 10 seconds a positive finding is recorded, and the number of positive sites is recorded and then expressed as a percentage of the number of the sites examined.

CONTACTS AND LOCATIONS:
Overall Officials: Merna N Elnahas, Master's degree, Principal Investigator — Mansoura Unniversity
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided